CLINICAL TRIAL: NCT07128914
Title: A Phase I Clinical Trial Evaluating the Safety, Tolerability, and Preliminary Efficacy of GO306 Recombinant Oncolytic Vaccinia Virus Injection in Patients With Advanced Refractory Solid Tumors.
Brief Title: A Clinical Study of GO306 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GeneSail Biotech (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-CN-GO306-202501
Record Dates: First submitted 2025-07-14; First posted 2025-08-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor Malignancies
Keywords: GO306; Solid tumor malignancies; Oncolytic Viral Therapy

STUDY DESIGN:
Intervention Model Description: This is a single-arm, non-randomized study which comprises two parts:
  * Part 1: A 3+3 single-dose escalation phase to determine the Maximum Tolerated Dose (MTD), Dose-Limiting Toxicities (DLTs), and Recommended Phase II Dose (RP2D) of the investigational product.
  * Part 2: A multiple-dose expansion phase at the RP2D level to explore preliminary efficacy in specific tumor types.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GO306 Treatment (Experimental): This is a single-arm, non-randomized study which comprises two parts:
  * Part 1: A 3+3 single-dose escalation phase to determine the Maximum Tolerated Dose (MTD), Dose-Limiting Toxicities (DLTs), and Recommended Phase II Dose (RP2D) of the investigational product.
  * Part 2: A multiple-dose expansion phase at the RP2D level to explore preliminary efficacy in specific tumor types.
  Interventions: Drug: GO306

INTERVENTIONS:
Drug: GO306 — Part 1: A 3+3 single-dose escalation phase:
  Low-dose cohort: 3.0E+07 PFU; Intratumoral or intracavitary injection of GO306; Cohort Size: 3 subjects; Dosing Schedule: Single initial administration.
  Medium-dose cohort: 3.0E+08 PFU; Intratumoral or intracavitary injection of GO306; Cohort Size: 3 subjects; Dosing Schedule: Single initial administration.
  High-dose cohort: 1.0E+09 PFU; Intratumoral or intracavitary injection of GO306; Cohort Size: 3 subjects; Dosing Schedule: Single initial administration.
  Part 2: A multiple-dose expansion phase at the RP2D level to explore preliminary efficacy in specific tumor type:
  RP2D; Intratumoral or intracavitary injection of GO306; Cohort Size: 20 subjects in specific tumor type; Dosing Schedule: QW or Q2W administration.

SUMMARY:
This study employs a single-arm, open-label, non-randomized, dose-escalation design to investigate the safety, tolerability, and efficacy of GO306 Recombinant Oncolytic Vaccinia Virus Injection.

* Part 1: Utilizes the 3+3 design principle to evaluate the safety and tolerability of a single administration of GO306 at different dose levels. The primary goal is to determine the Maximum Tolerated Dose (MTD), providing the basis for selecting the Recommended Phase 2 Dose (RP2D).
* Part 2: Evaluates the safety and tolerability of repeated intratumoral (IT) or intracavitary administrations of GO306 in patients with specific tumor types.

DETAILED DESCRIPTION:
This study employs a single-arm, open-label, non-randomized, dose-escalation design to investigate the safety, tolerability, and efficacy of GO306 Recombinant Oncolytic Vaccinia Virus Injection. The study has two parts.

* Part 1 is a single-dose escalation phase.

  * The Main Objectives of part 1 is to evaluate the safety and tolerability of single intratumoral injection/intracavitary administration of GO306 at different dose levels in patients with advanced solid tumors who failed to respond to standard treatment, and explore the maximum tolerated dose (MTD), so as to provide a basis for the recommended dose in the second stage.
  * The secondary objectives of Part 1 is 1) To evaluate the pharmacokinetics (PK) and viral shedding of GO306 after single intratumoral injection/intracavitary administration; 2) evaluate the preliminary efficacy of a single dose of GO306; 3) To monitor the changes of immunological parameters related to GO306 pharmacodynamics.
  * The exploratory objectives of Part 1 is to correlation between PD-L1 expression in tumor tissue, microsatellite instability (MSI), tumor mutation burden (TMB) and efficacy (if applicable);
* Part 2 Multiple dose exploration phase.

  * The primary objective of Part 2 is to evaluate the safety and tolerability of multiple intratumoral injection/intracavitary administration of GO306 in patients with specific tumors and to determine the optimal dosing regimen.
  * The secondary objectives of Part 2 is 1) To evaluate the pharmacokinetics (PK) and viral shedding of GO306 after multiple intratumoral injections/intracavitary administration; 2) evaluate the preliminary efficacy of multiple doses of GO306; 3) evaluate the immunogenicity of GO306; 4) To monitor the changes of immunological indicators related to GO306 pharmacodynamics.
  * The exploratory objectives of Part 2 is to correlation between PD-L1 expression in tumor tissue, microsatellite instability (MSI), tumor mutation burden (TMB) and efficacy (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old and above, regardless of gender.
* Patients with histologically or cytologically confirmed advanced malignant solid tumors, including but not limited to breast cancer, bladder urothelial cancer, colorectal cancer, renal cancer, ovarian epithelial cancer, and neuroendocrine tumors, who have no response or failure to standard treatment (including disease progression and/or intolerable side effects), or no standard treatment. Examples are as follows:

  * a. Histologically or cytologically confirmed unresectable or metastatic bladder urothelial carcinoma: failure to or intolerance to prior platinum-based chemotherapy and PD-1/PD-L1 inhibitors or no available standard treatment options for unresectable or metastatic disease.
  * b. Patients with histologically or cytologically confirmed recurrent ovarian cancer with malignant ascites who have received at least one previous line of platinum-based chemotherapy-based therapy and no available standard treatment options, and those with germline or somatic BRCA mutations who failed or did not tolerate PARP inhibitors.
  * c. Histologically or cytologically confirmed unresectable or metastatic colorectal cancer with liver metastases: failure or intolerance to prior oxaliplatin, fluorouracil, and irinotecan based therapy (or PD-1/PD-L1 inhibitors if the patient is MSI-H/dMMR) or no standard treatment options are available.
  * d. Patients with histologically or cytologically confirmed unresectable or metastatic clear-cell renal carcinoma with prior failure to, or intolerance to, Tkis and PD-1/PD-L1 inhibitors or no available standard treatment options for unresectable or metastatic clear-cell renal carcinoma.
  * e. Histologically or cytologically confirmed, locally advanced or metastatic triple-negative breast cancer: failure to or intolerance to at least one previous line of standard chemotherapy, which must include a taxane (e.g., paclitaxel, docetaxel), or no standard treatment options available.
  * f. For patients with neuroendocrine tumors, one of the following criteria must be met:

    * (1) Patients with histologically confirmed advanced stage (inoperable locally advanced or distant metastasis) with Ki-67≥55% in G3 NET and NEC (including mixed neuroendocrine and non-neuroendocrine tumors [at least 30% neuroendocrine carcinoma component], excluding small cell lung cancer and Meckel cell carcinoma) : They have failed or are intolerant to at least one previous line of standard chemotherapy (EP or EC), or no standard treatment options are available.
    * (2) Histologically confirmed advanced NET G3 patients (unresectable locally advanced or distant metastasis) and atypical pulmonary and mediastinal carcinoid patients: patients who had received at least second-line standard treatment failed or could not tolerate it, and the treatment regimen must include CAPTEM regimen or no available standard treatment regimen.
  * g. Histologically or cytologically confirmed advanced solid tumors (other than the above, e.g., soft tissue sarcoma, etc.) : documented disease progression or intolerance during or after receiving previous standard therapy, or no standard treatment options are available.
* Patients with ovarian cancer and solid malignant tumors of the digestive tract with malignant ascites who plan intracavitary injection should meet the following requirements:

  * a. Malignant ascites was pathologically diagnosed as caused by the spread of cancer cells.
  * b. Grade ≥2 ascites recurred within 4 weeks after receiving at least one local treatment (including paracentesis, intraperitoneal chemotherapy, intraperitoneal venous shunt, hyperthermic intraperitoneal perfusion, etc.).
  * c. Massive peritoneal effusion confirmed by computed tomography (CT) or B-ultrasound, which clinically requires local treatment for peritoneal effusion.
* At least one lesion that could be evaluated, as confirmed by local imaging, according to RECIST 1.1 criteria. Intratumoral injectable lesion, with or without CT/ ultrasound guidance, was defined as a palpable or CT/ ultrasound visible skin, subcutaneous, or deep mass with a major diameter ≥1.5cm (in the case of a lymph node, a short diameter ≥1.5cm) amenable to CT/ ultrasound guidance for intratumoral injection, as judged by the investigator. The injection site was required to have not been treated with radiation.
* Eastern Cooperative Oncology Group (ECOG) score ≤2.
* Expected survival time ≥3 months.
* The subjects had adequate organ function at the baseline of the screening period, and the laboratory indicators met the following criteria:

  * a. Hematopoietic system (no previous blood transfusion or hematopoietic stimulating factor therapy within 14 days) : absolute neutrophil count (ANC) ≥1.5×109/L; Hemoglobin (Hgb) ≥90g/L; Platelet count (Plt) ≥75×109/L.
  * b. Liver function: serum total bilirubin (TBIL) ≤1.5×ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN, with liver metastasis TBIL≤3×ULN, ALT and AST≤5×ULN; Serum albumin ≥2.8 g/dL (subjects could use albumin to meet criteria).
  * c. Renal function: serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (according to Cockroft-Gault formula) >50mL/min.
  * d. Coagulation: international normalized ratio (INR) ≤1.5, activated partial thromboplastin time (APTT) ≤1.5×ULN.
* Participants were willing and able to comply with protocol requirements for the duration of the trial, including but not limited to receiving treatment, using effective contraception (for 3 months after dose), and undergoing regular follow-up and examinations.

Exclusion Criteria:

* Female subjects who were pregnant or lactating.
* Patients who had received a diagnosis of another malignancy within the previous 2 years, except for cancers with a low risk of metastasis and death (5-year survival rate, >90%), such as adequately treated basal-cell or squamous-cell skin cancer or carcinoma in situ of the cervix and other cancers in situ.
* The adverse effects of previous antitumor treatment have not returned to CTCAE v5.0 grade 1, baseline or lower, or the level specified in the inclusion/exclusion criteria (except for alopecia, hyperpigmentation and other adverse events judged by the investigator as no safety risk). Subjects with chronic grade 2 toxicity were eligible after discussion with the sponsor if they were asymptomatic or adequately controlled with stable medications.
* Antineoplastic therapy, including chemotherapy, radiotherapy, biotherapy, endocrine therapy, or immunotherapy, was received within 4 weeks or five half-lived periods (whichever was less) before the first use of the investigational drug, except for the following drugs: nitrosourea or mitomycin C within 6 weeks before the first use of the investigational drug; For oral fluorouracil and small molecule targeted drugs, 2 weeks before the first use of the investigational drug or within the 5 half-lives of the drug, whichever is longer; The Chinese herbal medicine or Chinese patent medicine with anti-tumor indication was within 2 weeks before the first use of the investigational drug.
* Presence of any of the following infections or diseases:

  * a. Active hepatitis B (HbsAg positive and/or HbcAb positive with an HBV DNA test value greater than the upper limit of normal); Active hepatitis C (anti-HCV antibody positive for further HCV RNA positive).
  * b. A known history of immunodeficiency virus (HIV) disease or HIV antibody positive or active syphilis.
  * c. evidence of clinically significant immunodeficiency such as a primary immunodeficiency state such as severe combined immunodeficiency (SCID); Opportunistic bacterial infection.
* Have a history of active autoimmune disease requiring systemic therapy such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc., or have been receiving long-term systemic steroids (prednisone >10mg/ day or equivalent dose of the same drug) or any other form of immunosuppressive therapy within 14 days before the first use of the investigational drug. Patients with clinically stable autoimmune thyroid disease were excluded. The patients were treated with topical and inhaled corticosteroids, such as ocular, intra-articular, nasal, etc. Short-term use of glucocorticoids (not more than 3 days) for prophylaxis (e.g., to prevent contrast allergy); Physiological doses of hormone replacement therapy.
* Received allogeneic tissue or solid organ transplantation.
* A history of severe cardiovascular and cerebrovascular disease, including but not limited to:

  * a. New York Heart Association (NYHA) class ≥II congestive heart failure.
  * b. left ventricular ejection fraction (LVEF) <50%.
  * c. QT interval corrected with Fridericia's method (QTcF) >470 ms or syndrome of prolonged QT interval.
  * d. Acute coronary syndrome, aortic dissection, major arrhythmia, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months before the first dose of dose.
  * e. Presence of uncontrolled hypertension (systolic BP, >150 mmHg or diastolic BP, >100 mmHg) Subjects with a history of hypertension were allowed to participate if blood-pressure control below this criterion was achieved and maintained with antihypertensive treatment.
* Patients with grade 3 or above bleeding events in the previous 6 months; Or patients with > grade 2 bleeding, hemangioma/vascular malformation, tumor stroke, tumor invasion of blood vessels, active gastrointestinal ulcer, and esophageal varices, who were judged by the investigators to have a significant risk of bleeding.
* A history of severe skin disease requiring systemic treatment within the previous 2 years, such as eczema, atopic dermatitis, burns, seborrheic dermatitis, psoriasis, severe acne, etc.
* Patients with severe allergy or hypersensitivity reaction after using any drug or biological product in the past.
* Anticoagulants or antiplatelet drugs should be used before intratumoral injection and should not be interrupted, including aspirin within 7 days before injection; Coumarin that cannot be stopped within 7 days before injection; Direct thrombin inhibitors (e.g., dabigatran) or direct factor Xa inhibitors (e.g., rivaroxaban, apixaban and endoixaban) that cannot be stopped within 4 days before injection; "Low-molecular-weight heparin (e.g., low-molecular-weight heparin [LMWH]), which cannot be discontinued within 24 hours before injection, and unfractionated heparin (e.g., unfractionated heparin [UFH]), which cannot be discontinued more than 4 hours before injection."
* Use of systemic immunomodulatory drugs within 14 days before the first use of the investigational drug, including but not limited to thymosin, IL-2, IFN, etc.
* Other circumstances requiring systemic anti-infective treatment within 4 weeks prior to the first administration of the investigational product, including but not limited to hospitalization for infectious complications, bacteremia, severe pneumonia, or active tuberculosis.
* Within 4 weeks before the first use of the investigational drug: receiving other unmarketed investigational drugs or treatments, and receiving live vaccines or live attenuated vaccines.
* Subjects who had undergone major surgery requiring hospitalization within 4 weeks before the first use of the investigational drug, or who were expected to undergo major surgery during the trial.
* Concomitant use of sensitive substrate drugs metabolized by CYP450 enzymes with a narrow therapeutic window that cannot be stopped within the first 5 half-lives of the investigational drug is recommended after discussion with the sponsor.
* Any known mental illness or substance abuse that may interfere with the subject's ability to cooperate with the trial.
* According to the evaluation of the investigators, the treatment risks are high, including but not limited to the high risk of bleeding, possible damage to the surrounding important tissue structures, the risk of shock caused by dizzy with blood and needles, and the risk of aggravating local infection.
* If the participant plans to participate in another clinical trial during the trial period, plans to leave the trial site, or otherwise is not suitable for participation in the trial as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
AEs | Within 6 Months After the Last Treatment
  Adverse events (AEs) will be graded according to the CTCAE Version 5.0 published by the U.S. National Cancer Institute.
SAEs | Within 6 months after the last treatment.
  Severe Adverse events (SAEs) will be graded according to the CTCAE Version 5.0 published by the U.S. National Cancer Institute.
DLT | Up to 21 days from the first GO306 injection.
  The Dose-Limiting Toxicities (DLTs) assessed using the NCI CTCAE v5.0.
MTD | Up to 21 days from the first GO306 injection.
  The maximum tolerated dose (MTD) of GO306 will be defined based on the DLT
RP2D | Through the Part 1 of this study, an average of 4 months
  The Recommended Phase II Dose (RP2D) will be determined based on the integrated analysis of Part 1 (3+3 dose-escalation phase) results.

SECONDARY OUTCOMES:
Pharmacodynamics/immunological indicators | In Part 1&2: Within 28 Days After the Last Dose
  Including but not limited to: peripheral blood T lymphocyte subsets (CD3+, CD4+, CD8+, CD4+/CD8+ ratio, CD19+, etc.), plasma cytokines (IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, IL-17, IFN-α, IFN-γ, TNF-α, etc.)
Pharmacokinetics/viral shedding indicators | Part 1&2: Within 28 Days After the Last Dose
  GO306 concentration (viral genome copy number) in blood, throat swabs, urine, saliva, feces, and injection site samples at different time points after a single dose, and the concentration of GO306 expression products in serum
Immunogenicity indicators | Part 1&2: Within 6 Months After the Last Dose
  Anti-GO306 antibodies, and antibodies against GO306 expression products.
OS | Up to 5 years after the last treatment.
  Overall Survival (OS)(Basd on the RECIST V1.1): Time interval from the date of first study drug administration to the date of death due to any cause.
PFS | Up to 5 years after the last treatment.
  Progression-Free Survival (PFS)(Basd on the RECIST V1.1): Time from first dose to the earlier occurrence of disease progression per RECIST 1.1 or death from any cause.
ORR | Up to 5 years after the last treatment.
  Objective Response Rate (ORR)(Basd on the RECIST V1.1): Proportion of subjects achieving a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) per RECIST 1.1, assessed from first dose until treatment discontinuation.
DOR | Up to 5 years after the last treatment.
  Duration of Response (DOR)(Basd on the RECIST V1.1): Time from the first documented CR or PR until PD or death from any cause, whichever occurs first, as assessed per RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Shenzhen Third People's Hospital, Shenzhen, Guangzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shanghai General Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No